CLINICAL TRIAL: NCT06429176
Title: A Phase 2a, Randomized, Placebo-Controlled, Double Blind Multiple Ascending Dose Study in Patients with Cystic Fibrosis Carrying the 3849 +10 Kb C->T Mutation to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of SPL84
Brief Title: Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of SPL84 in Patients with Cystic Fibrosis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: SpliSense Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: SPL84-002; 2024-511184-28 (EudraCT Number)
Record Dates: First submitted 2024-05-15; First posted 2024-05-24 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-11

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- SPL84 (Active Comparator)
  Interventions: Drug: SPL84
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: SPL84 — SPL84 solution for nebulization
  Arms: SPL84
Other: Placebo — Placebo solution for nebulization
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if drug SPL84 is safe for adult patients with cystic fibrosis (CF). It will also learn if the drug works to treat works to treat CF with a specific mutation.

The purpose of this research study is to:

* test the safety and effectiveness of multiple doses of the study drug, SPL84
* test how multiple doses of the drug are processed by the body

Researchers will compare drug SPL84 to a placebo (a look-alike substance that contains no drug) to see if drug SPL84 is safe and if it works to treat CF.

Participants will:

Take drug SPL84 or a placebo by inhalation every week for 9 weeks months Visit the clinic approximately 14 times over 17.5 weeks for checkups and tests

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CF and two CF causing mutations; 3849+10 Kb C->T mutation on one allele in the CF transmembrane conductance regulator (CFTR) gene (homozygote or compound heterozygote). Source documentation from a certified genetic laboratory is required.
* Body mass index (BMI) of ≥ 17 kg/m2.
* FEV1 40-90% predicted at screening.
* Non-smokers or vapers for at least 180 days (6 months) prior to screening, per participant report.

Exclusion Criteria:

* Use of Kalydeco, Orkambi, Symdeko/Symkevi or Trikafta/Kaftrio within 30 days of first dose with study intervention.
* Use of any investigational drug (other than SPL84) or device within 30 days of first dose with study intervention.
* Use of systemic steroids over 3 consecutive months in the last 6 months prior to screening, or use of systemic steroids in the last month prior to screening. Use of inhaled steroids above 1 mg.
* Use of CF medications, e.g. inhaled antibiotics, dornase alfa (Pulmozyme), hypertonic saline and physiotherapy should be on stable regimen for the period 28 days prior to screening; those participants taking inhaled antibiotics for prophylaxis must be on a stable regimen of these drugs for at least 90 days prior to first dose with study intervention.
* Any acute infection including acute upper respiratory or lower respiratory infections, pulmonary exacerbation, changes in therapy for pulmonary disease, or any non CF-related illness which results in the initiation of any new therapy within 14 days prior to first dose with study intervention.
* Hemoptysis of greater than 30 mL within 90 days prior to Day 1, or hospitalization for hemoptysis within 6 months of first dose with study intervention.
* Liver disease characterized by clinically significant cirrhosis and/or documented portal hypertension.
* History of any organ transplantation.
* Documented coronavirus disease (COVID-19) infection within 4 weeks prior to dosing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability of SPL84 as evaluated by number of subjects with at least one treatment-related adverse event (AE) or serious adverse event (SAEs) | Day 1 through Day 87
  Incidence, nature, and severity of AEs and SAEs
Safety and Tolerability of SPL84 as assessed by number of participants with abnormal heart rate | Day 1 through Day 87
Safety and Tolerability of SPL84 as assessed by number of participants with abnormal respiratory rate | Day 1 through Day 87
Safety and Tolerability of SPL84 as assessed by number of participants with abnormal systolic and diastolic blood pressure | Day 1 through Day 87
Safety and Tolerability of SPL84 as assessed by number of participants with abnormal oximetry | Day 1 through Day 87
Safety and Tolerability of SPL84 as assessed by number of participants with abnormal temperature | Day 1 through Day 87
Safety and Tolerability of SPL84 as assessed by number of participants with abnormal hematology lab test results | Day 1 through Day 87
Safety and Tolerability of SPL84 as assessed by number of participants with abnormal biochemistry lab test results | Day 1 through Day 87
Safety and Tolerability of SPL84 as assessed by number of participants with abnormal urinalysis lab test results | Day 1 through Day 87
Safety and Tolerability of SPL84 as assessed by number of participants with abnormal electrocardiogram (ECG) parameters | Day 1 through Day 87
  using an ECG machine that automatically calculates heart rate and measure PR, QRS, QT, and QTc intervals
Safety and Tolerability of SPL84 as assessed by number of participants with abnormal physical examination findings | Day 1 through Day 87
  Complete physical examinations include general appearance, head, ears, eyes, nose, throat, thyroid, chest (heart, lungs), abdomen, skin, neurological, extremities, back, neck, musculoskeletal, and lymph nodes.
Safety and Tolerability of SPL84 as assessed by number of participants with abnormal pulmonary function tests results | Day 1 through Day 87
  Pulmonary function tests will be performed according to the American Thoracic Society (ATS)/European Respiratory Society (ERS) and forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC), and forced mid-expiratory flow (FEF25-75) will be measured
Safety and Tolerability of SPL84 as assessed by number of participants with abnormal sputum microbiology results results | Day 1 through Day 87
  Sputum microbiology will be performed with a microbiology based assay; organism growth will be identified.
Safety and Tolerability of SPL84 as assessed by number of participants with abnormal immunogenicity results | Day 1 through Day 87
  assessment of anti-SPL84 antibodies will be performed both in serum and sputum

SECONDARY OUTCOMES:
Characterization of pharmacokinetics (PK) of SPL84: maximum serum concentration (Cmax) | Predose and 15 and 30 minutes and 1, 2, 4, 6, 8, and 24 hours postdose on Day 1 and Day 57; predose on Days 8 and 29; Days 64 and 87
Characterization of PK of SPL84: Time to Cmax (Tmax) | Predose and 15 and 30 minutes and 1, 2, 4, 6, 8, and 24 hours postdose on Day 1 and Day 57; predose on Days 8 and 29; Days 64 and 87
Characterization of PK of SPL84: terminal elimination half-life (t1/2) | Predose and 15 and 30 minutes and 1, 2, 4, 6, 8, and 24 hours postdose on Day 1 and Day 57; predose on Days 8 and 29; Days 64 and 87
Characterization of PK of SPL84: Area under the curve to the final sample (AUC0-t) | Predose and 15 and 30 minutes and 1, 2, 4, 6, 8, and 24 hours postdose on Day 1 and Day 57; predose on Days 8 and 29; Days 64 and 87
Characterization of PK of SPL84: Area under the curve to infinity (AUC0-∞) | Predose and 15 and 30 minutes and 1, 2, 4, 6, 8, and 24 hours postdose on Day 1 and Day 57; predose on Days 8 and 29; Days 64 and 87
Characterization of PK of SPL84: Apparent clearance (CL/F) | Predose and 15 and 30 minutes and 1, 2, 4, 6, 8, and 24 hours postdose on Day 1 and Day 57; predose on Days 8 and 29; Days 64 and 87
Characterization of excretion of SPL84: concentration of SPL84 in urine | Day 1 through Day 87
Preliminary efficacy of SPL84 as assessed by change from baseline in percent predicted FEV1 | Day 1 through Day 87
  Pulmonary function tests will be performed according to the ATS/ERS
Preliminary efficacy of SPL84 as assessed by change from baseline in Cystic Fibrosis Questionnaire-Revised Respiratory Symptom Score | Day 1 through Day 87
  The score for is standardized on a 0- to 100-point scale on which higher scores represent a higher quality of life
Preliminary efficacy of SPL84 as assessed by change from baseline in body weight | Day 1 through Day 87
Preliminary efficacy of SPL84 as assessed by change from baseline of antibiotic treatment | Day 1 through Day 87

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Boston Children'S Hospital, Boston, Massachusetts
  - Nationwide Children'S Hospital, Columbus, Ohio